CLINICAL TRIAL: NCT01048359
Title: Multidisciplinary Approach to Reduce Injury and Substance Abuse
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DESPR DA026088; 5R01DA026088-02 (NIH)
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Drug Abuse
Keywords: Drug abuse, injury, trauma, screening, brief intervention.
MeSH Terms: conditions — Substance-Related Disorders; Wounds and Injuries | interventions — Crisis Intervention; Immunization, Secondary

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Brief Intervention (Experimental): 30-45 minute motivational interviewing based intervention with feedback addressing drug use, injury prevention and HIV risk.
  Interventions: Behavioral: Brief Intervention
- Brief advice (Active Comparator): This condition of the experiment acts a control and will be a short session in which the therapist will provide brief advice about drug use and give the patient a pamphlet.
  Interventions: Behavioral: Brief advice
- Brief Intervention plus Booster (Experimental): 30-45 minute motivational interviewing based intervention with feedback addressing drug use, injury prevention and HIV risk plus a brief phone booster session at 1 month post-intake to review feedback, 2) assess progress, 2) renew motivation to change, and 3) evaluate and affirm commitment to change.
  Interventions: Behavioral: Brief Intervention plus Booster

INTERVENTIONS:
Behavioral: Brief advice — The American College of Surgeons (ACS) recently mandated standards of care for all level I trauma centers and currently defined standards of care at the collaborating institution requires that assessment and referral are included in treatment as usual. Therefore, our treatment as usual, or BA, consists of an initial interview conducted by study staff, a recommendation to abstain from drug use, provision of educational material supporting that recommendation, referral to hospital or community treatment resources most likely to be beneficial to the patient and information about relevant community health care agencies.
  Arms: Brief advice
Behavioral: Brief Intervention plus Booster — A brief drug use intervention based on motivational interviewing is provided to participants at baseline and a booster session incorporating personalized feedback is provided at one month
  Arms: Brief Intervention plus Booster
Behavioral: Brief Intervention — A brief drug use intervention based on motivational interviewing is provided to participants at baseline
  Arms: Brief Intervention

SUMMARY:
The primary purpose of the project entitled: Multidisciplinary Approach to Reduce Injury and Substance Abuse, which is funded by the National Institute on Drug Abuse (5R01DA026088-02), is to compare the effectiveness of brief intervention, brief intervention plus a booster, and brief advice for adult patients who abuse drugs and present to a trauma department for treatment of an injury.

DETAILED DESCRIPTION:
Multidisciplinary Approach to Reduce Injury and Substance Abuse is a randomized clinical trial evaluating the effectiveness of brief advice (BA), brief motivational intervention with feedback (BMI), and brief motivational intervention with feedback and booster (BMI+B) in injured patients with drug problems.

The setting is a level 1 Trauma Department, which serves a large and diverse patient population. Injured patients are screened for eligibility in the project based on a positive toxicology screen or self reported drug use in the past 90 days. The primary outcome of interest will be patients' subsequent drug use. Other outcomes of interest include: HIV-related risk behaviors, improved health outcomes (including injury reduction), increased employment, decreased engagement in illegal behavior, increased substance abuse treatment utilization, and enhanced quality of life at three, six, and twelve month follow-ups.

This study will also examine the potential moderating and mediating effects of patient readiness to change, use of experiential and behavioral processes of change and decisional balance considerations. In addition, this project will examine implementation factors at the organizational level and the cost effectiveness of BA, BMI, and BMI+B.

Study participants and their related identifying information will be collected during the time they are admitted to the recruitment hospital trauma department. Study participants must be 18 years or older, speak English or Spanish, have been admitted to the recruitment hospital trauma department, and test positive for illegal drugs or admit to illegal drug use when verbally screened. Additional information will be collected from participants in the in-person assessment interviews at three, six, and 12 month follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must be 18 years or older
* Speak English or Spanish
* Been admitted to the level 1 Trauma Department
* Test positive for illegal drugs or admit to illegal drug use

Exclusion Criteria:

* Other penetrating trauma not related to motor vehicle collisions, violence or falls, such as poisoning and, bites
* Patients with traumatic brain injury, or a Glasgow Coma Scale score of less than 15
* Patients who do not pass the Mini-Mental Status Exam are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome of interest will be patients' subsequent drug use. | 3, 6, and 12 months after intervention

SECONDARY OUTCOMES:
HIV risk-behaviors, improved health, increased employment, decreased illegal behavior, increased substance treatment, enhanced quality of life, use of Transtheoretical model of change, organization implementation, and intervention cost-effectiveness. | 3, 6, and 12 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Velasquez, PhD, Principal Investigator — University of Texas at Austin; Craig A Field, PhD, Principal Investigator — University of Texas, El Paso
Locations (1):
- University Medical Center Brackenridge, Austin, Texas, United States